CLINICAL TRIAL: NCT04968379
Title: An Open-Label, Multi-Center Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Intravenous Ferric Carboxymaltose (FCM) in Infants (0-1 Year) With Iron Deficiency Anemia
Brief Title: Safety, Tolerability, PK and PD of Intravenous Ferric Carboxymaltose in Infants With Iron Deficiency Anemia
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficult to recruit and enroll patients for this study in a reasonable amount of time.
Sponsor: American Regent, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1VIT19046
Record Dates: First submitted 2020-11-02; First posted 2021-07-20 (Actual); Last update posted 2023-01-06 (Actual); Status verified 2023-01

CONDITIONS: Iron Deficiency, Anaemia
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — ferric carboxymaltose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ferric Carboxymaltose (Experimental): To evaluate the safety, tolerance, PK and PD profile of intravenous (IV) FCM in infants 0 to 1 year of age with IDA after receiving a 5.0 mg/kg dose of FCM
  Interventions: Drug: Ferric carboxymaltose
- Injectafer (Experimental): To evaluate the safety, tolerance, PK and PD profile of intravenous (IV) FCM in infants 0 to 1 year of age with IDA after receiving a 7.5 mg/kg dose dose of FCM.
  Interventions: Drug: Ferric carboxymaltose

INTERVENTIONS:
Drug: Ferric carboxymaltose — Intravenous
  Other Names: Injectafer

SUMMARY:
An Open-Label, Multi-Center Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Intravenous Ferric Carboxymaltose (FCM) in Infants (0-1 year) with Iron Deficiency Anemia.

DETAILED DESCRIPTION:
A phase II, open-label, multi-center study with 2 Cohorts to evaluate the safety, tolerance, PK, and PD profile of intravenous (IV) FCM in infants 0 to 1 year of age with IDA after receiving either a 5.0 mg/kg or 7.5 mg/kg dose of FCM.

Participants will have a screening evaluation within 14 days of the first dose of study drug. A medically supervised environment is required on Day 1 (day of dosing) and for 4 hours post dosing. Participants are allowed to be enrolled if satisfying the inclusion and exclusion criteria. Participants will return to the study site for additional evaluation and sampling on Days 8 (± 2 days), 15 (± 2 days), 22 (± 2 days), and 36 (± 2 days).

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants 0 to 1 year of age, medically indicated for iron replacement, with his/her parent or legal guardian willing and able to sign the informed consent form approved by the IRB / Independent Ethics Committee (IEC).
2. Screening Hb ≥7 g/dL to <10 g/dL.
3. Infants with any of the following conditions:

   * Heart failure with IDA defined as syndromes of excessive preload, excessive afterload, abnormal rhythm, or decreased contractility
   * Gastrointestinal diseases with acquired short bowel syndrome (due to volvulus, necrotizing enterocolitis from surgical resection or spontaneous intestinal perforation)
   * Gastrointestinal intolerance of oral iron or an unsatisfactory response to oral iron
   * Other conditions associated with IDA which in the opinion of the investigator might benefit from administration of FCM

Exclusion Criteria:

1. Known history of hypersensitivity reaction to FCM.
2. Body weight <2.5 kg.
3. History of acquired iron overload, hemochromatosis, or other iron accumulation disorders.
4. Hemodialysis-dependent chronic kidney disease.
5. History of significant diseases of the liver, hematopoietic system, cardiovascular system, or other conditions which, on the opinion of the investigator, may place a participant at added risk for participation in the study.
6. Active infection.
7. Anemia due to reasons other than iron deficiency (e.g., hemoglobinopathy vitamin B12 deficiency, or folic acid deficiency).
8. Blood transfusion in the 4 weeks prior to consent.
9. Administration of an iron-containing product within 14 days of administration of the study article.
10. Administration and / or use of an investigational product (drug or device) within 30 days of screening.
11. Current participation in another clinical trial.
12. Unable to comply with study procedures and assessments.

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2022-07-21 (Actual); Primary Completion 2024-10-08 (Estimated); Study Completion 2024-12-12 (Estimated)

PRIMARY OUTCOMES:
Treatment-emergent adverse events | Baseline to Day 36
  Treatment-emergent clinical laboratory test (clinical chemistry and hematology) abnormalities
Change in hemoglobin (Hb): g/dL | baseline to Days 8, 15, 22, and 36
  determine appropriate dosing of FCM in infants from 0 to 1 year of age by evaluating PD parameters
Change in reticulocytes count: % | baseline to Days 8, 15, 22, and 36
  determine appropriate dosing of FCM in infants from 0 to 1 year of age by evaluating PD parameters
Evaluate the PD parameters - Change in serum iron: mcg/dL | baseline to Day 36
  To determine appropriate dosing of FCM in infants from 0 to 1 year of age by evaluating PD parameters.
Evaluate the PD parameters - Change in serum ferritin: ng/mL | baseline to Day 36
  Description: To determine appropriate dosing of FCM in infants from 0 to 1 year of age by evaluating PD parameters.
Evaluate the PD parameters - Change in total iron binding capacity [TIBC]): mcg/dL | baseline to Day 36
  Description: To determine appropriate dosing of FCM in infants from 0 to 1 year of age by evaluating PD parameters.
Evaluate the PD parameters - Change in serum transferrin saturation [TSAT]): mg/dL | baseline to Day 36
  Description: To determine appropriate dosing of FCM in infants from 0 to 1 year of age by evaluating PD parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Falone, MD, Study Director — American Regent
Locations (4):
- United States (4):
  - University of Iowa, Iowa City, Iowa
  - Cohen Children's Medical Center, New Hyde Park, New York
  - Nationwide Children's Hospital, Columbus, Ohio
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania